CLINICAL TRIAL: NCT07139704
Title: The Effect of Mindfulness-Based Sexual Counseling on Body Appreciation, Sexual Distress, and Sexual Self-Confidence in Postpartum Women With Episiotomy
Acronym: Mindfulness-Ba
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Gul OZTAS, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIUIE7
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Women
Keywords: Mindfulness-Based Sexual Counseling; MİDWİFERY; Episiotomy; Postpartum Women; Body Appreciation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single (Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR-BA (Experimental): This study will aim to evaluate the effect of mindfulness-based sexual counseling on body appreciation, sexual distress, and sexual self-confidence in postpartum women with episiotomy.This randomized controlled experimental study will include participants assigned to intervention and control groups. The intervention group will receive a four-week mindfulness-based sexual counseling program consisting of eight sessions, while the control group will receive routine care. Body Appreciation, Sexual Distress, and Sexual Self-Confidence scales will be administered as pre- and post-tests.
  Interventions: Behavioral: Mindfulness-Based Sexual Counseling (MBSR-BA)
- control: (No Intervention): Routine Postpartum Care

INTERVENTIONS:
Behavioral: Mindfulness-Based Sexual Counseling (MBSR-BA) — A MBSR-based sexual counseling program applied to women after episiotomy, 2 sessions per week for 4 weeks, 8 sessions in total.
  Arms: MBSR-BA

SUMMARY:
Aim: This study will aim to evaluate the effect of mindfulness-based sexual counseling on body appreciation, sexual distress, and sexual self-confidence in postpartum women with episiotomy.

Method: This randomized controlled experimental study will include participants assigned to intervention and control groups. The intervention group will receive a four-week mindfulness-based sexual counseling program consisting of eight sessions, while the control group will receive routine care. Body Appreciation, Sexual Distress, and Sexual Self-Confidence scales will be administered as pre- and post-tests.

DETAILED DESCRIPTION:
An episiotomy is a surgical incision made in the perineal muscles during labor to widen the vaginal opening, facilitate the safe and rapid delivery of the fetal head, shorten the second stage, reduce the risk of lacerations, and prevent anal sphincter damage (Carroli & Mignini, 2009; Shmueli et al., 2017; Goh, Goh, & Ellepola, 2018; Deyaso et al., 2022). This intervention, normally recommended only for medical indications, has become routine in many countries over time. This has led international health authorities such as the World Health Organization (WHO), the American College of Obstetricians and Gynecologists (ACOG), and NICE to issue clear warnings against unnecessary episiotomy (WHO, 2018; ACOG, 2006; NICE, 2023; Ghulmiyyah et al., 2022). According to the WHO's 2018 guidelines, episiotomy rates vary widely between countries. In Southeast Asia, this rate reaches 63%, while in Europe the average is 20-25%. In Turkey, the overall rate is reported as 52%, 93.3% in primiparous women, and 30.2% in multiparous women. Similarly high rates are reported in developing countries such as India (63.4%), Oman (66%), Cambodia (94.5%), and Taiwan (100%) (Djusad et al., 2024). Episiotomy can affect women's health not only during labor but also in the postpartum period. Research shows that this intervention is associated with complications such as postpartum perineal pain, dyspareunia, decreased sexual desire, and orgasmic disorders (Dedavid da Rocha & Zamberlan, 2018; Khajehei et al., 2015; Buhling et al., 2018). Furthermore, episiotomy can cause sexual dysfunction, distorted body image, decreased sexual self-confidence, and lowered self-esteem (Khajehei et al., 2015; Buhling et al., 2018; Ghulmiyyah et al., 2022). Female sexual dysfunction is a condition characterized by lack of sexual desire, difficulty with arousal, orgasmic problems, and pain, which negatively affects an individual's quality of sexual life and psychological well-being. Its prevalence in the first 2-3 months after birth varies between 41-83% (De Souza et al., 2015). These disorders threaten psychological health by causing negative changes in body image and self-esteem (Ören & Yaşar, 2023; Naisri, 2015).

Mindfulness is a mind-body practice that allows individuals to focus on the present moment and observe thoughts, emotions, and bodily sensations without judgment (Durna et al., 2019). Regular practice increases levels of happiness, psychological flexibility, compassion, and self-compassion, and reduces levels of depression, anxiety, and stress (İnci & Ergen, 2019; Cengizhan & Uçar, 2023). The literature reports that mindfulness-based interventions have positive effects on sexual dysfunction, body image, and self-esteem. However, studies examining the effects of mindfulness-based sexual counseling on sexual distress, body image, and sexual self-confidence in postpartum women who have undergone an episiotomy are extremely limited. In societies where sexuality is considered taboo, such as those in southeastern Turkey, such an intervention is anticipated to provide benefits at both the individual and societal levels. This study aims to evaluate the effects of mindfulness-based sexual counseling on body image, sexual distress, and sexual self-confidence in postpartum women experiencing episiotomy. The study is expected to fill a gap in the literature and offer a holistic, evidence-based, and culturally sensitive intervention model for postpartum sexual health.

ELIGIBILITY:
Inclusion Criteria:

* Having had a vaginal birth and an episiotomy,

  * Having a follow-up appointment with the Family Health and Medical Center at 8 weeks postpartum,
  * Being able to read and write in Turkish,
  * Having a 3rd or 4th degree perineal tear

Exclusion Criteria:

* • History of pelvic surgery,

  * Significant psychiatric illness,
  * Presence of chronic illness that may affect sexual function

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — POSTPORTUM WOMEN
Enrollment: 124 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Distress Inventory-Revised (FSSI-R): | 4 WEEEK
  Developed by Derogatis et al. (2008) and adapted to Turkish by Aydın et al. (2016), it is a 13-item, five-point Likert-type scale assessing personal distress associated with sexual dysfunction. Possible scores range from 0 to 52, with higher scores indicating greater sexual distress. The cut-off point is ≥ 11.5. The Cronbach's alpha coefficient is 0.98.
Sexual Self-Esteem Scale (SSS) | 4 WEEK
  Developed by Çelik (2012), it consists of 13 items. Items are scored from 1 ("never") to 4 ("always"). The total score ranges from 13 to 52, with higher scores indicating higher sexual self-confidence. The Cronbach's alpha coefficient is 0.88.
Body Esteem Scale (BSS) | 4 WEEK
  Developed by Cragun (2013) and adapted to Turkish by Arslan et al. (2020). It is a 15-item, five-point Likert-type scale consisting of three subscales: body esteem-weight, body esteem-appearance, and body esteem-quality. The subscale Cronbach's alpha coefficients are 0.940, 0.920, and 0.810, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmama Universty, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No